CLINICAL TRIAL: NCT04100551
Title: Relationship Between Chronic Renal Disease Gradation and Risk Stratification for Chronic Ulcer on the on the Diabetic Foot
Brief Title: Relationship Between Chronic Renal Disease and Risk Stratification for Chronic Ulcer on the on the Diabetic Foot
Acronym: NEPHROPOD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0431
Record Dates: First submitted 2019-09-13; First posted 2019-09-24 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic Renal Disease; Diabetic Foot
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Context and hypothesis: The prevalence of diabetes mellitus keeps going to increase, due to the ageing of the population and the high prevalence of overweight and obesity. Thus about 5% of the French population is said to have diabetes according to the national health insurance reimbursement data estimations. 15 to 20% of diabetic patients will have a foot chronic ulcer in their lifetime. Nowadays, diabetes is still the leading cause of non-traumatic amputation in France, amputation being very often preceded by a trophic disorder. Thus, the person with diabetes has a 7-fold risk of amputation. For the year 2013, in France, incidence rates of hospitalizations for lower limb amputations and foot wounds in the diabetic population were 252/100000 and 668/100000 respectively. In an attempt to prevent the risk of foot wounds in people with diabetes, the International Working Group on the Diabetic Foot (IWGDF) has established foot grades associated with an increased risk of foot wounds. These grades are now used by health authorities to calibrate their care offer such as reimbursements for podiatry care. Chronic kidney disease is one of the major complications of diabetes. In 2013, according to data from the French registry (REIN), 4,856 diabetics started renal replacement therapy in 2016, representing 46% of the newly dialyzed population. This represents a relative risk 9.2 times higher than in the general population. The Investigators hypothesize that beyond the risk of wound, there is a link between the stage of chronic renal disease and the risk of foot ulcer grade as defined by the IWGDF. The link between chronic renal disease and this common marker of foot risk has never been studied to our knowledge. The long-term objective, beyond this study, is to improve patient pathways and thus improve the prevention of foot wounds in diabetics with renal insufficiency. This is all the more true since prevention actions in the dialysis population have already shown their effectiveness on a large scale on the risk of amputation.

Protocol : All patients with a diabetes mellitus who consult diabetology and nephrology services at the Montpellier University Hospital will be included in this study. The consultation wil be the same as usual. The Investigators will ask for the history of diabetes, the history of complications, the current treatments and the Investigators will make a standardized clinical examination of feet with a foot risk gradation according to the IWGDF.The investigators will report the standard biologicals values.

DETAILED DESCRIPTION:
A simple standardization of the clinical examination (Foot Risk Grading), history collection and biological data will be organized by the study sponsors.

List of collected data, origin and circuit of the data:

Entry of patient data (clinical, biological and additional examinations) on a database registered at the University Hospital of Montpellier on a secure server.

Data from :

* Computerized medical records and consultation letters.
* The question form completed by the physician- The results of biological examinations carried out outside or inside the university hospital vested with a standardized standard prescription form

All the data corresponds to the current annual or infra-annual follow-up of patients consulting for the pathologies studied: Diabetes and renal failure.

The data will be anonymized by a chronic search entry number and 1st letter of the surname and first name.

The statistical analysis of the data will be carried out internally at the Montpellier University Hospital, in collaboration with the Medical Information Department, in accordance with the partnerships already in place between our teams.

Data :

Simple demographic characteristics: Age, gender Clinical history: Longstanding diabetes, diabetic retinopathy, diabetic maculopathy, ischemic heart disease, history of stroke, lower limb arteriopathy, known gastroparesis, high blood pressure, hypercholesterolemia, microalbuminuria or known proteinuria.

Clinical features: BMI, lower limb neuropathy - monofilament test error, pulse abolition

. Treatments: diabetes, type of kidney substitution, other treatments Toxic: Tobacco, Alcohol Quality of patient follow-up: date of last ophthalmic consultation (For each diabetic person: one consultation per year is recommended - this criterion is monitored by health insurance as a quality criterion for follow-up)

Biological assessment: Creatinemia, Calcaemia, Phosphatemia, Magnesemia, 1.25OHVitD, 25OHVitD, 25OHVitD, Natremia, Kalemia, Albuminaemia, PTH, CRP, Uric acid, HbA1C, Hemoglobinaemia, HDL, LDL, Triglyceridaemia, Cholesterol, Albuminuria/Creatinuria ratio, Proteinuria/Creatinuria ratio

ELIGIBILITY:
Inclusion criteria:

* Diabetes type 1 or 2
* Consultation in nephrology or diabetology at the Montpellier university hospital

Exclusion criteria:

* Solid Organ transplant
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Diabetes type 1 or type 2 over 18 years old from the consultation of Diabetology or nephrology at the Montpellier university hospital
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
relationship between renal function and podological grade | 1 day
  Gradation of the Risk stratification for chronic ulcer on the diabetic foot by the IWGDF Chronic renal disease gradation with the Enzymatic measure of creatininemia. Clearance calculation with CKD-EPI. (CKD-EPI >90 ; 60-90 ; 45-60 ; 30-45 ; 15-30 ; < 15 ; Dialysis)

SECONDARY OUTCOMES:
factors associated with the occurrence of complications and comorbidities | 1 day
  Cardiovascular disease
factors associated with the occurrence of complications and comorbidities | 1 day
  current biological rates
factors associated with the occurrence of complications and comorbidities | 1 day
  HbA1C

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC